CLINICAL TRIAL: NCT00456885
Title: The Effect of Exenatide on Body Weight, Energy Expenditure and Hunger in Obese Women Without Diabetes Mellitus
Brief Title: The Effect of Exenatide on Weight and Hunger in Obese, Healthy Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Eleftheria Maratos-Flier, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2006P000361; BFA912
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Obesity; Impaired Glucose Tolerance
Keywords: obesity; double blind; placebo controlled; weight loss; appetite; energy expenditure
MeSH Terms: conditions — Obesity; Glucose Intolerance; Weight Loss | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide First (Placebo Comparator): Started on Exenatide, 3 week washout, start placebo
  Interventions: Drug: exenatide; Drug: Placebo
- Placebo First (Experimental): Started on placebo, 3 week washout, start exenatide
  Interventions: Drug: exenatide; Drug: Placebo

INTERVENTIONS:
Drug: exenatide — 5 microgram twice a day for two week and then 10 mcg for remaining 15 weeks
  Other Names: Byetta
Drug: Placebo — Twice daily injection of placebo

SUMMARY:
This study will look at the effect of exenatide, a drug which has been approved for the treatment of type 2 diabetes, on body weight, appetite and energy expenditure among moderately obese women without diabetes.

The study is 35 weeks long and includes 19 outpatient visits. Participants will receive exenatide for 16 weeks and placebo for 16 weeks with a 3 week rest period in between. Neither participants nor investigators will know whether exenatide or placebo is being administered. Participants will be started randomly on either exenatide or placebo.

Our hypothesis is that treatment with exenatide will curb appetite and lead to weight loss and may lead to changes in energy expenditure.

DETAILED DESCRIPTION:
This study will examine the effect of exenatide on body weight, energy expenditure, satiety, sleep, and metabolic parameters in healthy, moderately obese women (BMI 28-35 kg/m2). We will look at 2 populations of women, one with normal glucose metabolism and one with impaired glucose homeostasis (IGH)--either impaired fasting glucose (IFG, fasting glucose 101-125 mg/dL) or impaired glucose tolerance (IGT, glucose 140-199 mg/dL 2h after a 75g oral glucose load). This is a randomized, double blind, crossover study with two 16-week treatment periods separated by a 3-week washout period. There are 19 study visits over 35 weeks.

The goals of this study are 1) to examine the effect of exenatide on body weight and dysglycemia in populations in which this medication has not been studied, namely obese women with and without IGH and 2) to investigate possible mechanisms of weight loss through measurements of energy expenditure, hunger, satiety, nausea, and sleep.

The primary outcome of this study is weight loss. We will calculate absolute and relative change in body weight from baseline to week 16 (the first treatment period) and from week 19 to week 35 (the second treatment period). Body weight will be measured at every study visit which will also allow us to assess the absolute and relative change from baseline throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 25-60
2. BMI 28-35 kg/m2
3. No known diagnosis of diabetes
4. No known diagnosis of coronary heart disease
5. Self-described sedentary lifestyle with minimal regular cardiovascular exercise (no more than 1 hour per week)
6. Stable weight (variation < 3 kg within 6 months of screening visit)
7. Ability to give informed consent
8. Ability to follow verbal and written instructions
9. Use of medically approved form of contraception (monophasic oral contraception, intra uterine device, surgical sterilization or 2 combined barrier methods)
10. Nonsmoker (tobacco, marijuana)
11. Outpatient visits every 2 weeks throughout the study period are required. While most of these visits are short (15 minutes)ability to commute to the performance site in Boston, on a regular basis, is necessary.

Exclusion Criteria:

1. Type 1 or type 2 diabetes mellitus diagnosed according to American Diabetes Association criteria
2. Coronary heart disease (history of myocardial infarction or unstable angina pectoris)
3. Uncontrolled hypertension hypertension (BP > 150/90 mmHg on or off antihypertensive medication)
4. Uncontrolled dyslipidemia (LDL > 200 or TG > 400 on or off lipid lowering medication)
5. Tobacco, marijuana or intravenous drug use
6. Shift workers (night shift or alternating day/night shifts)
7. Recent weight loss (> 3 kg within 4 months of the screening visit)
8. Gastroparesis
9. Inflammatory bowel disease
10. Malignancy treated with chemotherapy within the past 3 years
11. History of pancreatitis
12. Depression requiring hospitalization or diagnosis of psychosis
13. Renal insufficiency (creatinine clearance < 50 ml/min)
14. Transaminases > 2x above the normal range
15. Pregnancy within 6 months of the screening visit
16. Breastfeeding
17. Failure to use medically approved contraceptive methods
18. History of an eating disorder (anorexia, bulimia or laxative abuse)
19. History of surgery for the treatment of obesity (gastric banding, gastric bypass, gastric stapling)
20. New diagnosis of hypo or hyperthyroidism within 1 year of screening visit
21. Previous participation in a clinical study with exenatide
22. Presence or history of allergic reaction to multiple drugs

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleftheria Maratos-Flier, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Dushay J, Gao C, Gopalakrishnan GS, Crawley M, Mitten EK, Wilker E, Mullington J, Maratos-Flier E. Short-term exenatide treatment leads to significant weight loss in a subset of obese women without diabetes. Diabetes Care. 2012 Jan;35(1):4-11. doi: 10.2337/dc11-0931. Epub 2011 Oct 31. PMID 22040840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Flyers, Craig's list, posters used for recruitment.Recruitment occurred between 2007 and 2010. After telephone screen subjects were evaluated at the BIDMC clinical research center.
Groups:
- Exenatide First, Then Placebo: Started on exenatide, 3 week washout, started on placebo.
- Placebo First, Then Exenatide: Started on placebo, three week washout, started on exenatide.
Period: First Treatment Period, 16 Weeks
Arm/Group | Exenatide First, Then Placebo | Placebo First, Then Exenatide
Started | 24 | 17
Completed | 24 | 17
Not Completed | 0 | 0
Period: Washout, 3 Weeks
Arm/Group | Exenatide First, Then Placebo | Placebo First, Then Exenatide
Started | 24 | 17
Completed | 24 | 17
Not Completed | 0 | 0
Period: Second Treatment Period, 16 Weeks
Arm/Group | Exenatide First, Then Placebo | Placebo First, Then Exenatide
Started | 24 | 17
Completed | 23 | 17
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants in the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 41
Weight [Mean (Standard Deviation); unit: Kilograms] | 89 (14)
BMI [Mean (Standard Deviation); unit: Kg/meter^2] | 33 (4)
HOMA IR [Mean (Standard Deviation); unit: Ratio] — This is the ratio of fasting glucose to fasting insulin. It has no definable upper limit. We are showing scores in our study participants.
  Ratio | 2 (1)
Waist [Mean (Standard Deviation); unit: centrimeters] — centimeters
  centrimeters | 105 (12)
Body Fat [Mean (Standard Deviation); unit: percent] — Measured using bio-electrical impedance
  percent | 40 (5)
Systolic BP [Mean (Standard Deviation); unit: mm of mercury] | 128 (14)
Diastolic BP [Mean (Standard Deviation); unit: mm of Mercury] | 75 (8)
HDL [Mean (Standard Deviation); unit: mg/dl] | 62 (19)
LDL [Mean (Standard Deviation); unit: mg/dl] | 114 (28)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 198 (32)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 111 (64)
Fasting Insulin [Mean (Standard Deviation); unit: mU per liter] | 8 (6)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dl] | 85 (12)
Two Hour Glucose [Mean (Standard Deviation); unit: mg/dl] | 110 (32)
Adiponectin [Mean (Standard Deviation); unit: micrograms/ml] | 6 (3)
Leptin [Mean (Standard Deviation); unit: ng/ml] | 36 (18)
Resting Energy Expenditure [Mean (Standard Deviation); unit: Kilocalories] — Using indirect calorimetry
  Kilocalories | 1439 (196)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Change in weight at the end of each treatment period.
Time Frame: 16 weeks after the beginning of each treatment
Measure: Mean (Standard Error); unit: kilograms
Groups:
- Exenatide: All participants that received exenatide.
- Placebo: All participants that received placebo.
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
kilograms | -2.49 (0.66) | 0.43 (0.63)

2. Primary Outcome: Change in Body Mass Index
Time Frame: 16 weeks from the start of each treatment period.
Measure: Mean (95% Confidence Interval); unit: Kg/m^2
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
Kg/m^2 | -0.93 [-1.44 to -0.41] | 0.18 [-0.31 to 0.68]

3. Secondary Outcome: Change in Waist Circumference
Time Frame: 16 weeks from the start of each treatment period.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
centimeters | -1.68 [-3.3 to -0.07] | 0.94 [-0.59 to 2.47]

4. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure was measured using a Dynamap automated monitoring device. The change is reported as the blood pressure measured at the beginning of the treatment group and after 16 weeks. We are reporting the change in the systolic blood presssure recorded.
Time Frame: 16 weeks after the beginning of each treatment
Measure: Mean (95% Confidence Interval); unit: mm of mercury
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
mm of mercury | -2.5 [-6.6 to 1.6] | -1.3 [-5.2 to 2.6]

5. Secondary Outcome: Changes in Body Composition
Description: Per cent body body fat was assessed using bio-electrical impedance with a BIA; RJL System Quantum II Bioelectrical Body Composition Analyzer. The data is reported as per cent body fat.
Time Frame: 16 weeks after the beginning of each treatment
Measure: Mean (95% Confidence Interval); unit: per cent
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
per cent | -0.4 [-1.5 to 0.7] | -0.7 [-1.8 to 0.3]

6. Secondary Outcome: Changes in Leptin
Time Frame: 16 weeks from the start of each treatment period.
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
ng/ml | -3.7 [-7.4 to 0.05] | -0.2 [-3.8 to 3.3]

7. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 16 weeks after the beginning of each treatment
Measure: Mean (95% Confidence Interval); unit: mm of mercury
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
mm of mercury | -1.2 [-3.6 to 1.1] | -0.4 [-2.6 to 1.9]

8. Secondary Outcome: Adiponectin
Time Frame: 16 weeks after the beginning of each treatment
Measure: Mean (95% Confidence Interval); unit: microgram per ml
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
microgram per ml | 0.4 [-0.3 to 1.0] | 0.07 [-0.5 to 0.7]

9. Secondary Outcome: Change in Insulin
Time Frame: 16 weeks from the start of each treatment period.
Measure: Mean (95% Confidence Interval); unit: microunits per liter
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
microunits per liter | 1.1 [-0.6 to 2.8] | 0.4 [-1.3 to 2.0]

10. Secondary Outcome: Change in Fasting Glucose
Time Frame: 16 weeks from the start of each treatment period.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
mg/dl | 0.5 [-3.6 to 4.5] | 3.1 [-0.7 to 7.0]

11. Secondary Outcome: Change in Two Hour Glucose
Time Frame: 16 weeks from the start of each treatment period.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
mg/dl | -10 [-21 to 1.2] | -0.5 [-11 to 10]

12. Secondary Outcome: HOMA Score
Time Frame: 16 weeks from the start of each treatment period.
Measure: Mean (95% Confidence Interval); unit: Ratio fasting glucose to insulin
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
Ratio fasting glucose to insulin | 0.2 [-0.3 to 0.6] | 0.2 [-0.3 to 0.6]

13. Secondary Outcome: REE
Description: Resting Energy Expenditure
Time Frame: 16 weeks from the start of each treatment period.
Measure: Mean (95% Confidence Interval); unit: Kilocalories
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 41 | 40
Kilocalories | -13.7 [-60.6 to 33.2] | 6.5 [-38.0 to 51.0]

ADVERSE EVENTS:
Time Frame: 37 weeks
Description: Adverse effects were monitored as all participant adverse events and were not monitored by intervention or sequence.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 31/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=41)
Nausea (Gastrointestinal disorders) | 31 — Nausea
Bloating (Gastrointestinal disorders) | 1 (1) — Bloating
Irritation at injection site (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No